CLINICAL TRIAL: NCT06990464
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SIBP-A19 Injection in the Treatment of Advanced Malignant Solid Tumor Patients
Brief Title: A Clinical Trial of SIBP-A19 Injection in the Treatment of Advanced Malignant Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-A19-I
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumor; ADC; Safety; Efficacy; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This study is an open, multicenter, dose escalation, dose expansion, and indication expansion study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIBP-A19 (Experimental): The participants enrolled will be sequentially assigned to the corresponding dose level.
  Interventions: Drug: SIBP-A19

INTERVENTIONS:
Drug: SIBP-A19 — SIBP-A19 formulation for injection. Strength: 1.0, 2.0, 3.2, 4.0, 4.8, 5.6, 6.4 and 8.0 mg/kg. Intravenous infusion administration, with a treatment cycle of every 21 days, administered once on the first day of each cycle. The dose escalation stage, 1mg/kg and 2mg/ kg were subjected to accelerated titration, where the safety was evaluated within 21 days after the first administration to one participant. If dose-limiting toxicity (DLT) occurred, the traditional "3+3" dose escalation method was immediately switched. If DLT does not occur, the next dose group will be explored. The third stage will use RP2D for further exploration.

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetic characteristics of SIBP-A19 and determine the maximum tolerable dose (MTD) and phase II recommended dose (RP2D).

DETAILED DESCRIPTION:
This study is an open label, multicenter, dose escalation, dose expansion, and indication expansion study to evaluate safety, tolerability, pharmacokinetics, preliminary anti-tumor efficacy, immunogenicity, impact on QT/QTc interval, and explore potential biomarkers of SIBP-A19 for injection in participants with advanced or metastatic solid tumors.

This study is divided into three stages and is planned to be set up eight dose groups, including 1.0, 2.0, 3.2, 4.0, 4.8, 5.6, 6.4 and 8.0 mg/kg. The first stage is the dose escalation stage, which will start from the first and second doses for enrollment. If necessary, a 3+3 dose escalation design will be used. The second stage is the dose expansion stage, where two or more doses are selected to enter the dose expansion phase, and 6-9 participants will be enrolled in each dose group for dose expansion. The third stage is the indication expansion stage, where phase II recommended dose (RP2D) is preliminarily determined based on the escalation and expansion of dosage in the early stage. Using RP2D for indication expansion, the investigators plan to expand three indication cohorts, with at least 30 participants selected for each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 75 years old (including boundary values), regardless of gender.
* Voluntarily participate in this study and sign the informed consent form.
* Participants with advanced or metastatic solid tumors diagnosed by histology or cytology, without standard treatment, standard treatment failure, or intolerance.
* Willing and able to provide sufficient fresh collected or archived tumor tissue samples or provide testing reports from legitimate institutions that meet the requirements.
* There must be at least one measurable lesion as the target lesion.
* ECOG score 0-1.
* Expected survival time ≥ 3 months.
* During the screening period, the main organ functions were basically normal (no medical support such as blood transfusion, granulocyte colony-stimulating factor (G-CSF), or other medical support was received within 14 days before the use of the investigational drug):

  • Blood routine: Absolute value of neutrophils (NE #) ≥ 1.5 × 10 9/L, platelet (PLT) count

  ≥ 90 × 10 9/L, hemoglobin (HGB) ≥ 90 g/L.
* Women of childbearing age during the screening period who have a negative blood pregnancy test and are capable of reproduction (including male participants) have no pregnancy plan and voluntarily take effective contraceptive measures during the trial period and within 6 months after the last dose.

Exclusion Criteria:

* Participants with the following tumors:

  * The participant has had other malignant tumors that have not been cured within the past 5 years (excluding malignant tumors that have been clearly cured, such as thyroid cancer, cured basal cell carcinoma of the skin, and cervical carcinoma in situ).
  * The participant has untreated imaging confirmed central nervous system metastasis.
  * Meningeal metastases.
  * Patients with brain metastases who have received systematic or curative brain metastasis treatment (radiotherapy or surgery) in the past, have been confirmed stable by imaging for at least 4 weeks, and have stopped systemic hormone, antiepileptic, convulsive drugs, and other treatments for more than 2 weeks without clinical symptoms can be enrolled.
* Participants with a history of previous treatment or surgery, or those who received the following anti-tumor treatments during the planned trial period:

  * Patients who accepted the instructions clearly containing traditional Chinese patent medicines and simple preparations with anti-tumor effect within 2 weeks before the first administration;
  * Patients undergoing adjuvant therapy within 6 months after surgery;
  * Patients who have not recovered from the toxicity of the previous anti-tumor treatment to normal or ≤ level 1 (excluding hair loss);
  * Patients who have undergone major surgery, radiation therapy, biological therapy, or chemotherapy within 4 weeks prior to their first administration, or who have received systemic treatment such as unhealed surgical wounds, ulcers or fractures, or other clinical trial drugs.
  * Patients who plan to receive any other anti-tumor treatment (chemotherapy, radiation therapy, immunotherapy, cytokine therapy other than erythropoietin) during the trial period should be excluded (excluding testosterone lowering therapy for prostate cancer patients).
  * The dose (prednisone>10 mg/d or equivalent) at which immunosuppressive effects are achieved by receiving immunosuppressive agents or systemic corticosteroids within one week prior to the use of the investigational drug.
* Participants with a history of previous illnesses or laboratory tests that show the following abnormalities:

  * Individuals with abnormal coagulation function and a tendency to bleed, or who are undergoing thrombolysis or anticoagulation treatment or have lost blood or donated more than 400 mL within 2 months prior to administration.
  * Have a history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
  * Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia.
  * Known history of drug abuse, alcoholism, or drug use that may affect the results of the trial.
* According to the investigator's judgment, the screening period is accompanied by serious, progressive, or uncontrolled diseases, and the investigator's assessment determines that the participant's participation in the study will increase the risk.
* According to the investigator's judgment, there are serious accompanying diseases that pose a threat to patient safety or affect the completion of the study.
* Patients with uncontrolled ascites, pleural effusion, pericardial effusion during the screening period or those who require drainage, or those who have undergone serosal fluid drainage within 4 weeks before the first administration.
* Patients who must take supplements containing folic acid (such as those with folate deficiency).
* Individuals with a history of severe allergies to protein products, CHO cell products, other recombinant human or humanized antibodies, or components of the investigational drug.
* Pregnant and lactating women.
* Patients who are deemed unsuitable to participate in this clinical study due to other reasons by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
AE (Adverse Events) | From day 1 after the first dose to day 28 after the last dose
  That is adverse events, any adverse events that occurred to the participant during the study period.
Phase II recommended dose (RP2D) | Day 21 after the last dose in the dose expansion phase
  RP2D refers to the recommended dose determined through initial dose escalation and toxicity assessment in clinical trials, used for further evaluation of drug efficacy and safety.
Dose-limiting toxicity (DLT) | Day 21 after each dose in the dose escalation stage
  DLT is defined as any adverse event related to the drug defined in the protocol that occurs within 21 days of the first cycle after a single administration.
Maximum tolerated dose (MTD) | Day 21 after the last dose in the dose escalation stage
  MTD is defined as the maximum dose at which the number of DLT cases occurring during the DLT observation period within 21 days after a single administration is ≤ 1/6 of the total number of cases.

SECONDARY OUTCOMES:
AUC (Area Under The Plasma Concentration Versus Time Curve) | Day 1, Day 22 and Day 63 after the first dose
  It shows the degree to which a drug is absorbed and used in the body.
Cmax (Peak Plasma Concentration) | Day 1, Day 22 and Day 63 after the first dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax (Peak Time) | Day 1, Day 22 and Day 63 after the first dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the participant plasma concentration curve after administration.
ORR (Objective Response Rate) | 6 weeks after the last evaluation
  The proportion of participants whose tumor volume shrinks to a predetermined value and maintains the minimum time limit and is the sum of complete and partial responses.
DCR (Disease control rate) | 6 weeks after the last evaluation
  In clinical trials, the percentage of participants with advanced cancer who responded fully to cancer treatment, partially responded, and had stable disease.
PFS (Progression-free survival) | 6 weeks after the last evaluation
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
OS (overall survival) | 6 weeks after the last evaluation
  From randomization to time of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ling ying Wu, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- The Union Hospital affiliated to Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No